CLINICAL TRIAL: NCT03245541
Title: A Phase I/II Study of Durvalumab (Medi 4736) and Stereotactic Ablative Body Radiotherapy in Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Radiation Therapy in Combination With Durvalumab for People With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-228
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Stereotactic Ablative Body Radiotherapy (SABR); Durvalumab; 20-228
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + SABR (Experimental): Durvalumab + Stereotactic Ablative Body Radiotherapy
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Ablative Body Radiotherapy (SABR)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be given 750 mg, intravenously (IV) over 60 minutes (+/- 5 minutes), Q14 days beginning D1. Four doses of durvalumab will be administered on the Q14 day schedule. Subsequently Durvalumab will continue as maintenance 1500mg, intravenously (IV) over 60 minutes (+/- 5 minutes), Q28 days up to 1 year or until progression (11 doses), unacceptable toxicity or other reason. If a patient undergoes resection, they will resume durvalumab once appropriately healed from surgery (approximately 4-8 weeks) at discretion of treating medical oncologist.
  Other Names: Medi 4736
Radiation: Stereotactic Ablative Body Radiotherapy (SABR) — SABR delivered as 6.6 Gy/fraction x 5 fractions given within two weeks will be administered weekdays and will begin D8.

SUMMARY:
The purpose of this study is to find out if combining durvalumab with standard stereotactic ablative radiotherapy (SABR) is an effective treatment for people with locally advanced or borderline resectable pancreatic cancer. The researchers will also look at the safety of the combination treatment and any side effects it causes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologic or cytologic diagnosis of adenocarcinoma of the pancreas (PDAC), or suspicious for malignancy per pathology, which is deemed BR or LA PDAC per NCCN guidelines or following evaluation by a Multidisciplinary group of physicians.
* Patients must have received FOLFIRINOX for 3-6 months prior to enrollment with at least stable disease by restaging imaging.

Note: SOC treatment regimen derived from FOLFIRINOX dose modifications are acceptable.

To maximize potential efficacy no more than a 6-week treatment break is recommended between the completion of SOC chemotherapy (FOLFIRINOX) and initiation of study treatment (durvalumab).

* Age ≥ 18 years
* Body weight >30kg
* ECOG 0-2
* Patients must have normal organ and marrow function as defined below:

  * Absolute Neutrophil Count (ANC) ≥1.0 K/mcL
  * Platelets ≥75 K/mcL
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤ 2.5 X ULN
  * Creatinine OR creatinine clearance ≤ 1.5 times the upper limit of normal OR > 40 mL/min for patients with creatinine levels above normal.

Note: Patients with biliary stent are eligible provided that all other inclusion criteria are met.

* Negative pregnancy test in women of childbearing potential (WOCBP) within 30 days of durvalumab administration or evidence of post-menopausal status. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Non-sterilized male participants who are sexually active with a female partner of childbearing potential must be willing to use a highly effective method of contraception from Day 1 through 90 days after receipt of the final dose of investigational product(s). Not engaging in sexual activity for the total duration of the study and the drug washout period is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male participants must be willing to refrain from sperm donation throughout these periods.
* Ability to understand and the willingness to sign an informed consent document.
* Willingness and ability to comply with the protocol including study treatment, scheduled assessments and follow-up.

Exclusion Criteria:

* History of another primary malignancy except for:

  °Malignancy treated with curative intent with no known active disease for 2 years before the first dose of study drug and low potential risk for recurrence.
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Patients who have had prior anti-cancer treatment or are currently receiving anti-cancer treatment for their disease other than chemotherapy as stipulated by protocol.
* Women who are breastfeeding.
* Any clinically significant, unresolved toxicity >CTCAE grade 2 from previous anti-cancer therapy with the exception of alopecia, vitiligo and laboratory values defined in the inclusion criteria.
* Patients with Grade ≥ 2 neuropathy will be included at the investigator's discretion
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included at the nvestigator's discretion
* Patients who are currently receiving any other investigational agents for therapeutic treatment of their primary cancer.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including Durvalumab or other immunotherapy.
* Known metastatic disease.
* Major surgical procedures based on clinical judgement of the investigator within 30 days prior to the first dose of study drug. Patients may undergo staging laparoscopy, PTC placement, ERCP, etc. at any time which should not interfere with study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are receiving radiation treatment outside of the enrolling centers.
* Patients with frank transmural macroscopic invasion of duodenum by tumor as determined by treating investigator.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis, Crohn's disease], diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel syndrome, or other serious gastrointestinal chronic conditions associated with diarrhea); systemic lupus erythematosus; Wegener syndrome (granulomatosis with polyangiitis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis, etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion: Patients with vitiligo or alopecia. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement, or psoriasis not requiring systemic treatment
* Current or prior use of immunosuppressive medication within 28 days before treatment, except with chemotherapy.
* History of organ transplant that requires use of immunosuppressive agents.
* History of active primary immunodeficiency.
* Receipt of live attenuated vaccination within 30 days prior to receiving durvalumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings and TB testing in line with local practices), active bleeding diatheses, hepatitis B (known positive HBV surface antigen result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).
* Patient with known active Hepatitis (i.e. Hepatitis B or C).

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg and PCR negative) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Patients with macroscopic invasion of the bowel or stomach submucosa by primary pancreatic tumor as determined by PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities in the first 10 weeks of treatment | 10 weeks
Progression Free Survival | 12 months
  Duration of time from diagnosis to time of progression
Proportion of participants who have resectable disease | 24 weeks
  Based on overall downstaging of disease post-treatment
Progression Free Survival (Phase II) | 6 months
  From study enrollment to time of progression

SECONDARY OUTCOMES:
Mean change in levels of inflammatory cytokines from baseline | 10 weeks
  As measured from cytokine analysis from serum
Mean change in levels of immune cells from baseline | 10 weeks
  As determined from flow cytometry from biopsies and blood
Mean change in protein levels from baseline | 10 weeks
  As determined from quantitative immunohistochemistry on biopsy samples
Mean change in microbiome from baseline | 10 weeks
  As determined from analysis of stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm